CLINICAL TRIAL: NCT03615066
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Safety, Tolerability and Antiviral Activity of GS-9688 in Viremic Adult Subjects With Chronic Hepatitis B Who Are Not Currently on Treatment
Brief Title: Study to Evaluate the Safety, Tolerability, and Antiviral Activity of Selgantolimod (Formerly GS-9688) in Viremic Adult Participants With Chronic Hepatitis B (CHB) Who Are Not Currently on Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-389-2025
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — selgantolimod; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Selgantolimod 3 mg + TAF (Experimental): Participants with Hepatitis B e antigen (HBeAg)-positive CHB or HBeAg-negative CHB currently not on oral antiviral (OAV) treatment, will receive selgantolimod 3 mg (2 x 1.5 mg tablet) on the same day once weekly for 24 doses along with tenofovir alafenamide (TAF) 25 mg once daily for 24 weeks. After the 24th dose, selgantolimod will be discontinued, and participants will continue to receive TAF until Week 48/early discontinuation (ED). At Week 48, per Principal Investigator's (PI's) discretion, participants can continue in the Treatment Free Follow-Up (TFFU) phase for up to an additional 48 weeks.
  Interventions: Drug: Selgantolimod; Drug: TAF
- Selgantolimod 1.5 mg + TAF (Experimental): Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, will receive selgantolimod 1.5 mg (1 x 1.5 mg tablet) and placebo (1 tablet) on the same day once weekly for 24 doses along with TAF 25 mg once daily for 24 weeks. After the 24th dose, selgantolimod will be discontinued, and participants will continue to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Placebo; Drug: Selgantolimod; Drug: TAF
- Placebo + TAF (Placebo Comparator): Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, will receive 2 tablets of placebo on the same day once weekly for 24 doses along with TAF 25 mg once daily for 24 weeks. After the 24th dose, placebo will be discontinued, and participants will continue to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Placebo; Drug: TAF

INTERVENTIONS:
Drug: Placebo — Tablet(s) administered orally every 7 days for 24 doses in fasted state
  Arms: Placebo + TAF; Selgantolimod 1.5 mg + TAF
Drug: Selgantolimod — Tablet(s) administered orally every 7 days for 24 doses in fasted state
  Other Names: GS-9688
  Arms: Selgantolimod 1.5 mg + TAF; Selgantolimod 3 mg + TAF
Drug: TAF — Tablet(s) administered orally once daily with food
  Other Names: Vemlidy®

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of multiple oral doses of selgantolimod and to evaluate the antiviral activity of selgantolimod in adult participants with chronic hepatitis B (CHB) who are viremic and not currently being treated.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Adult male and non-pregnant, non-lactating females
* Documented evidence of chronic hepatitis B virus (HBV) infection with detectable hepatitis B surface antigen (HBsAg) levels at screening
* Screening HBV deoxyribonucleic acid (DNA) ≥ 2000 international units per milliliter (IU/mL).
* Screening electrocardiogram (ECG) without clinically significant abnormalities

Key Exclusion Criteria:

* Extensive bridging fibrosis or cirrhosis
* Received a commercially available HBV OAV treatment(s) within the 3 months prior to screening.
* Received prolonged therapy with immunomodulators or biologics within 3 months of screening
* Individuals meeting any of the following laboratory parameters at screening:

  * Alanine aminotransferase > 5 * upper limit of normal (ULN)
  * International normalized ratio > ULN unless the individual is stable on an anticoagulant regimen
  * Albumin < 3.5 g/dL
  * Direct bilirubin >1.5x ULN
  * Platelet Count < 100,000/µL
  * Estimated creatinine clearance < 60 mL/min (using the Cockcroft-Gault method)
* Co-infection with human immunodeficiency virus (HIV), hepatitis C virus or hepatitis D virus
* Prior history of hepatocellular carcinoma or screening alpha-fetoprotein ≥ 50 ng/mL without imaging
* Diagnosis of autoimmune disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease, hemoglobinopathy, retinal disease, or are immunosuppressed.
* Chronic liver disease of a non-HBV etiology except for non-alcoholic fatty liver disease.
* Received solid organ or bone marrow transplant.
* Use of another investigational agent within 90 days of screening, unless allowed by the sponsor.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- Canada (3):
  - University of Calgary Liver Unit - Heritage Medical Research Clinic, Calgary, Alberta
  - University Health Network, Toronto General Hospital, Toronto Centre for Liver Disease, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen D, Kim S, Brooks A, McDonald C, Yang J, Gaggar A, et al. Potential Biomarkers of Response in Chronic Hepatitis B Patients Who Achieved HBeAg Loss Upon Treatment With Toll-Like Receptor 8 Agonist Selgantolimod [Poster]. The Digital International Liver Conference 2020 27-29 August.
- [Background] Janssen H, Lampertico P, Chen C-Y, Heo J, Foumier C, Ahn S, et al. Safety and Efficacy of Switching to Tenofovir Alafenamide in Virally Suppressed Chronic Hepatitis B Patients With Renal Impairment: Week-48 Results From a Phase 2 Open-label Study [Poster]. The Digital International Liver Conference 2020 27-29 August.
- [Background] Janssen H, Lim Y-S, Kim HJ, Tseng C-H, Coffin C, Elkashab M, et al. Safety and Efficacy of Oral TLR8 Agonist Selgantolimod in Viremic Adult Patients With Chronic Hepatitis B [Poster]. International Liver Congress 2021 23-26 June.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada, South Korea, and Taiwan. The first participant was screened on 28 August 2018. The last study visit occurred on 12 April 2021.
Pre-assignment Details: 96 participants were screened.
Groups:
- Selgantolimod 3 mg + TAF: Participants with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B (CHB) or HBeAg-negative CHB currently not on oral antiviral (OAV) treatment, received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses along with the tenofovir alafenamide (TAF) 25 mg orally once daily for 24 weeks. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/early discontinuation (ED). At Week 48, per Principal Investigator's (PI's) discretion, participants can continue in the Treatment Free Follow-Up (TFFU) phase for up to an additional 48 weeks.
- Selgantolimod 1.5 mg + TAF: Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, received selgantolimod 1.5 mg (1 x 1.5 mg tablet) and placebo (1 tablet) orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
- Placebo + TAF: Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, placebo was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
Period: Main Study
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Started | 26 | 28 | 13
Completed | 26 (2 participants did not receive all doses of study treatments but were considered to have completed the Main Study because the participants entered the TFFU Phase.) | 27 (1 participant did not receive all doses of study treatments but was considered to have completed the Main Study because the participant entered the TFFU Phase.) | 11
Not Completed | 0 | 1 | 2
Not completed — Withdrew Consent | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Treatment-free Follow-up (TFFU) Phase
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Started | 13 (13 participants who completed Main study did not enter TFFU phase.) | 12 (15 participants who completed Main study did not enter TFFU phase.) | 2 (9 participants who completed Main study did not enter TFFU phase.)
Completed | 11 | 11 | 2
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Groups:
- Selgantolimod 3 mg + TAF: Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF | Total
Number analyzed (Participants) | 26 | 28 | 13 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10.3) | 44 (12.1) | 46 (12.0) | 45 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 4 | 28
  Male | 15 | 15 | 9 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 27 | 13 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 25 | 28 | 13 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 15 | 6 | 33
  South Korea | 7 | 10 | 1 | 18
  Taiwan | 7 | 3 | 6 | 16
HBsAg [Mean (Standard Deviation); unit: log10 IU/mL] | 3.8 (0.86) | 4.2 (0.83) | 4.0 (0.73) | 4.0 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum Quantitative Hepatitis B Surface Antigen (qHBsAg) From Baseline at Week 24
Time Frame: Baseline, Week 24
Population: The Full Analysis Set included all randomized participants who took at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE was any unfavorable and unintended sign, symptom, disease, and/or laboratory or physiological observation that may or may not be related to the investigational medicinal product. A TEAE was defined as any AE with an onset date on or after the first dose date and no later than 30 days after permanent discontinuation of selgantolimod/placebo; or any AE leading to premature discontinuation of study drugs.
Time Frame: First dose date up to Week 24 plus 30 days
Population: The Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Groups:
- Selgantolimod 1.5 mg + TAF: Participants with HBeAg-positive CHB or HBeAg-negative CHB currently not on OAV treatment, received selgantolimod 1.5 mg (1 x 1.5 mg tablet) and placebo (1 tablet) orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 doses. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 84.6 | 60.7 | 76.9

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of the last dose of study drug plus 30 days for selgantolimod/placebo at Week 24. If the relevant baseline laboratory value was missing, any abnormality of at least Grade 1 observed within the time frame specified above was considered treatment emergent. Clinical laboratory results were graded according to Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities.
Time Frame: First dose date up to Week 24 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 84.6 | 92.9 | 92.3

4. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 4
Time Frame: Baseline, Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 8
Time Frame: Baseline, Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 12
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 4
Time Frame: Baseline, Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 25 | 27 | 13
log10 IU/mL | -0.04 (0.155) | -0.01 (0.081) | -0.02 (0.065)

9. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 8
Time Frame: Baseline, Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 23 | 28 | 12
log10 IU/mL | -0.04 (0.161) | -0.05 (0.121) | 0.00 (0.081)

10. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 12
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 27 | 12
log10 IU/mL | -0.04 (0.163) | -0.05 (0.108) | 0.01 (0.099)

11. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 28 | 12
log10 IU/mL | -0.08 (0.198) | -0.11 (0.174) | -0.03 (0.146)

12. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 27 | 11
log10 IU/mL | -0.12 (0.218) | -0.16 (0.235) | -0.12 (0.145)

13. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) < Lower Limit of Quantification (LLOQ) at Week 12
Description: LLOQ was defined as 20 IU/mL.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 28 | 12
percentage of participants | 20.8 | 28.6 | 25.0

14. Secondary Outcome: Percentage of Participants With HBV DNA < LLOQ at Week 24
Description: LLOQ was defined as 20 IU/mL.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 28 | 12
percentage of participants | 37.5 | 32.1 | 33.3

15. Secondary Outcome: Percentage of Participants With HBV DNA < LLOQ at Week 48
Description: LLOQ was defined as 20 IU/mL.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 27 | 11
percentage of participants | 50.0 | 44.4 | 45.5

16. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 12
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 25 | 28 | 12
percentage of participants | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 24
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 28 | 12
percentage of participants | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 48
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 24 | 27 | 11
percentage of participants | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 12
Description: HBeAg loss was defined as qualitative HBeAg changing from positive at baseline to negative at a postbaseline visit. HBeAg seroconversion was defined as Hepatitis B e antibody (HBeAb) loss and anti-HBe change from negative/missing at baseline to positive at a postbaseline visit.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed. Analysis was performed only on HBeAg-positive CHB participants.
Measure: Number; unit: percentage of participants
Groups:
- Selgantolimod 3 mg + TAF: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB currently not on OAV treatment, received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
- Selgantolimod 1.5 mg + TAF: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB currently not on OAV treatment, received selgantolimod 1.5 mg (1 x 1.5 mg tablet) and placebo (1 tablet) orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, selgantolimod was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
- Placebo + TAF: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB currently not on OAV treatment, received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses along with the TAF 25 mg orally once daily for 24 weeks. After the 24th dose, placebo was discontinued, and participants continued to receive TAF until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
Arm/Group | Selgantolimod 3 mg + TAF: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg + TAF: HBeAg-positive CHB Participants | Placebo + TAF: HBeAg-positive CHB Participants
Number analyzed (Participants) | 14 | 17 | 7
percentage of participants
  HBeAg Loss | 0 | 0 | 0
  HBeAg Loss and Seroconversion: number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 24
Description: HBeAg loss was defined as qualitative HBeAg changing from positive at baseline to negative at a postbaseline visit. HBeAg seroconversion was defined as HBeAb loss and anti-HBe change from negative/missing at baseline to positive at a postbaseline visit.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed. Analysis was performed only on HBeAg-positive CHB participants.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg + TAF: HBeAg-positive CHB Participants | Placebo + TAF: HBeAg-positive CHB Participants
Number analyzed (Participants) | 14 | 18 | 7
percentage of participants
  HBeAg Loss | 0 | 0 | 0
  HBeAg Loss and Seroconversion: number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 48
Description: HBeAg loss was defined as qualitative HBeAg changing from positive at baseline to negative at a postbaseline visit. HBeAg seroconversion was defined as HBeAb test changing from negative or missing at baseline to positive at a postbaseline visit.
Time Frame: Week 48
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg + TAF: HBeAg-positive CHB Participants | Placebo + TAF: HBeAg-positive CHB Participants
Number analyzed (Participants) | 14 | 17 | 6
percentage of participants
  HBeAg Loss | 0 | 0 | 0
  HBeAg Loss and Seroconversion: number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Virologic Breakthrough From Baseline up to Week 24
Description: Virologic breakthrough was defined as confirmed HBV DNA ≥ 69 IU/mL after having been < 69 IU/mL or confirmed HBV DNA ≥ 1 log10 IU/mL increase from nadir.
Time Frame: Baseline up to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 3.8 | 7.1 | 15.4

23. Secondary Outcome: Percentage of Participants With Virologic Breakthrough From Baseline up to Week 48
Description: as for outcome 22
Time Frame: Baseline up to Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 3.8 | 10.7 | 15.4

24. Secondary Outcome: Percentage of Participants With Drug Resistance Mutations
Time Frame: Baseline up to Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
Number analyzed (Participants) | 26 | 28 | 13
percentage of participants | 0 | 0 | 0

25. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Selgantolimod
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set (all randomized participants who took at least 1 dose of the study drug, participated in the optional intensive PK substudy, and had at least 1 nonmissing postdose concentration) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
hr*pg/mL
  Day 1 | 1163.0 (833.27) | 548.0 (393.00)
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 1441.8 (1601.19) | 491.2 (489.29)

26. Secondary Outcome: PK Parameter: AUC0-24 of Selgantolimod
Description: AUC0-24 is defined as the concentration of drug over time from time zero to time 24 hours.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
hr*pg/mL
  Day 1 | 1162.2 (832.29) | 547.7 (392.77)
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 1440.5 (1598.05) | 494.4 (485.56)

27. Secondary Outcome: PK Parameter: AUCinf of Selgantolimod
Description: AUC0-inf is defined as the concentration of drug over time from time zero to infinity.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
hr*pg/mL
  Day 1 | 1184.2 (843.53) | 556.4 (394.38)
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 1462.8 (1616.70) | 503.2 (492.66)

28. Secondary Outcome: PK Parameter: Cmax of Selgantolimod
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
pg/mL
  Day 1 | 373.3 (208.63) | 307.7 (311.12)
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 591.0 (565.11) | 268.2 (254.16)

29. Secondary Outcome: PK Parameter: Tmax of Selgantolimod
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
hours
  Day 1 | 0.98 [0.50 to 4.10] | 0.53 [0.28 to 1.80]
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 0.55 [0.28 to 1.10] | 0.50 [0.28 to 0.55]

30. Secondary Outcome: PK Parameter: CL/F of Selgantolimod
Description: CL/F is defined as the apparent oral clearance following administration of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
mL/hr
  Day 1 | 4094330.4 (3034917.79) | 4603039.8 (3733427.89)
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 4550308.6 (3858788.24) | 6223868.1 (5265428.49)

31. Secondary Outcome: PK Parameter: t1/2 of Selgantolimod
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours postdose at Day 1 and Week 23
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF
Number analyzed (Participants) | 7 | 8
hours
  Day 1 | 4.55 [4.32 to 4.95] | 5.13 [4.29 to 5.47]
  Week 23: number analyzed (Participants) | 3 | 5
  Week 23 | 4.78 [3.95 to 4.95] | 5.03 [4.76 to 5.10]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to Week 96 Adverse Events: First dose up to last dose of selgantolimod/placebo (Week 24) plus 30 days; or TAF (Week 48) plus 3 days, whichever came later
Description: All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse Events: The Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Arm/Group | Selgantolimod 3 mg + TAF | Selgantolimod 1.5 mg + TAF | Placebo + TAF
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/28 | 0/13
Other Adverse Events (participants affected / at risk) | 21/26 | 15/28 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selgantolimod 3 mg + TAF (N=26) | Selgantolimod 1.5 mg + TAF (N=28) | Placebo + TAF (N=13)
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selgantolimod 3 mg + TAF (N=26) | Selgantolimod 1.5 mg + TAF (N=28) | Placebo + TAF (N=13)
Palpitations (Cardiac disorders) | 3 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 6 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 0
Chest discomfort (General disorders) | 2 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 4 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 0
Feeling cold (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1 | 0
Headache (Nervous system disorders) | 3 | 5 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03615066/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03615066/SAP_001.pdf